CLINICAL TRIAL: NCT02029846
Title: Glycemia in Diabetic Elders Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No sufficient numbers of eligible participants
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00052707
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; Metformin; Sulfonylurea Compounds; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment (Active Comparator): A regimen with traditional drugs only
  Interventions: Drug: Standard Treatment
- Incretin-based Treatment (Experimental): A regimen including incretin-based drugs
  Interventions: Drug: Incretin-Based Treatment

INTERVENTIONS:
Drug: Standard Treatment — traditional drugs only
  Other Names: insulin; metformin; sulfonylureas; TZDs
  Arms: Standard Treatment
Drug: Incretin-Based Treatment — incretin-based drugs
  Other Names: GLP-1 analogues and receptor agonists,; DPP-4 inhibitors,; amylin analogues
  Arms: Incretin-based Treatment

SUMMARY:
This study is a pilot randomized controlled trial of 30 elderly type 2 diabetes patients conducted at the MODEL Clinical Research (MODEL), Research Division of Bay West Endocrinology Associates in Baltimore, Maryland. The investigators hypothesized that compared to a regimen base solely on traditional drugs, a regimen including newer drugs will achieve glycemic target faster and induce less hypoglycemia, weight gain, and other side effects, over the short run.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics diagnosed for at least 6 months
* Patients ages ≥ 65 years and older
* Active patients in the Bay West Endocrinology practice
* Inadequately controlled on oral agents and/or basal insulin with HbA1c between 8.0% and 12%
* Eligible for randomization to either treatment group
* Patients willing to follow either treatment arm including regimen using one or more injectables
* Patients to have an English Reading Level of Grade 6 or above
* Patients residing at home

Exclusion Criteria:

* Unwilling to use a regimen that may contain using one or more injections
* Using short acting insulin prior to the study
* Using GLP-1 in past 10 weeks
* History of hypoglycemia unawareness or episodes needing emergency intervention
* End-stage renal disease
* Dementia
* Blindness
* Terminal illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Chieh Yeh, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Bay West Endocrinology Associates, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment: A regimen with traditional drugs only
  Standard Treatment (insulin, metformin, sulfonylureas, TZDs): traditional drugs only
- Incretin-based Treatment: A regimen including incretin-based drugs
  Incretin-Based Treatment (GLP-1, DPP-4, amylin analogues): incretin-based drugs
Period: Overall Study
Arm/Group | Standard Treatment | Incretin-based Treatment
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — n=1 each arm | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Incretin-based Treatment | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 78 [78 to 78] | 67 [67 to 67] | 72.5 [67 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Glycemic Target (HbA1c <7.5%).
Description: Data not analyzed due to n=1 each arm.
Time Frame: 6 months
Population: Data not analyzed due to n=1 each arm.
Arm/Group | Standard Treatment | Incretin-based Treatment
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Hypoglycemia Measured by Glucose Meter
Description: Data not analyzed due to n=1 each arm.
Time Frame: 6 months
Population: Data not analyzed due to n=1 each arm.
Arm/Group | Standard Treatment | Incretin-based Treatment
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Diabetes Quality of Life
Description: Data not analyzed due to n=1 each arm
Time Frame: 6 months
Population: Data not analyzed due to n=1 each arm
Arm/Group | Standard Treatment | Incretin-based Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard Treatment | Incretin-based Treatment
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02029846/Prot_SAP_000.pdf